CLINICAL TRIAL: NCT05091463
Title: Non-invasive Spinal Stimulation as an Adjuvant Therapy for Trunk Control After Pediatric Spinal Cord Injury
Brief Title: Non-invasive Spinal Stimulation as an Adjuvant Therapy for Trunk Control After Pediatric SCI
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: The Craig H. Neilsen Foundation (Other)
Responsible Party: Principal Investigator, Andrea L. Behrman, PhD, PT, Professor, University of Louisville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21.0303
Record Dates: First submitted 2021-08-13; First posted 2021-10-25 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Spinal Cord Injuries
Keywords: Pediatric-onset; Transcutaneous spinal stimulation; Trunk deficit
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Transcutaneous spinal stimulation (Experimental): Participants with chronic SCI will receive 60 sessions of activity based-locomotor training (AB-LT) combined with transcutaneous stimulation (scTS).
  Interventions: Device: Biostim-5/Neostim transcutaneous spinal stimulator

INTERVENTIONS:
Device: Biostim-5/Neostim transcutaneous spinal stimulator — Transcutaneous spinal stimulation (scTS): The 5-channel stimulator capable of generating pain-free biphasic rectangular waveform of 0.3 to 1.0 ms pulses with a frequency of 5-10 kHz will be used to stimulate at single or multi-site spinal levels. Transcutaneous stimulation will be delivered in combination with activity based locomotor training in 5-10 minute bouts of stimulation at sub-motor threshold during daily sessions (5x/week) lasting for 90 minutes for a total of 60 sessions of therapy. The sessions will consist of 55-60 minutes on the treadmill for facilitated standing/stepping followed by 30 minutes of activities off the treadmill in sitting, standing, or stepping.

SUMMARY:
The overall purpose of this study is to test the efficacy of multi-modal training combining activity-based locomotor training and transcutaneous spinal stimulation (ABLT+scTS) to improve sitting posture and trunk control in children with a chronic spinal cord injury.

The investigators will recruit 12 participants, ages 3-12 with chronic, acquired SCI, T10 and above and non-ambulatory. The participants in this study will be novices to scTS and AB-LT.

DETAILED DESCRIPTION:
This is a within subjects, repeated measures design study. Participants with chronic, acquired SCI (T10 and above and non-ambulatory), ages 3-12 years will serve as their own control and will participate in the studies for all three aims. The participants in this study will be novices to scTS and AB-LT. Medical history and demographics will be collected according to NINDS-Common Data Elements guidelines for pediatric SCI and recommended, standardized outcomes used.

The participants will participate in 60 sessions, 5 days/week for 90 minutes/session. The participants will be assessed at the following time points: Baseline (prior to intervention), after 20 sessions, after 40 sessions and after 60 sessions.

If possible, there will be follow-up assessments occur at 3 months post-60 sessions.

Aim 1: To determine the effects of 60 AB-LT + scTS therapy sessions on sitting posture and trunk control.

Participants will be tested over a total of 4 session (2 pre- and 2 post-60 session intervention). Sessions 1 and 2 will include testing for clinical (Segmental Assessment of Trunk Control (SATCo) and Modified Functional Reach (MFR)) and biomechanical outcomes (Sitting with best posture and MFR), respectively. The two sessions will be conducted within one week.

Aim 2: Determine a) the rate of change in sitting posture and trunk control across, 20, 40, and 60 sessions of AB-LT + scTS, b) the durability of training effects at 3-months follow-up, and c) responsiveness of clinical outcome measures (SATCo and MFR) of trunk control.

Aim 3: To determine residual activation of trunk muscle below the level of the lesion, functional neurophysiological assessment (FNPA) and trunk perturbations will be assess pre- and post-intervention.

The investigators will attain parent/guardian informed consent and participant assent for children > 7 years. Twelve total participants, ages 3-12 years will be recruited and enrolled for all three aims. Participants will be enrolled for 60 sessions (3 months) for the intervention and will be re-tested 3 months post-training.

ELIGIBILITY:
Inclusion Criteria:

* Chronic (> 1 year since injury), Acquired Upper motor Neuron injury (T10 and above)
* Discharged from in-patient rehabilitation
* Moderate to severe trunk control deficit as assessed by the Segmental Assessment of Trunk Control (SATCo, score <16/20) OR unable to fully sit upright while lifting their arms or reaching outside of their base of support while maintaining posture
* Novice to activity-based locomotor training and transcutaneous spinal stimulation

Exclusion Criteria:

* Botox use within the past 3 months
* Current oral baclofen use and unwillingness or unable to wean under medical guidance
* Baclofen pump use
* Musculoskeletal impairment limiting range of motion, unhealed fracture, or other medical complication limiting participation
* Prior surgery for scoliosis
* Unwillingness to wean from the use of thoraco-lumbosacral orthosis (TLSO) during study
* Spina Bifida as etiology of spinal cord injury

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2021-08-31 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Segmental Assessment of Trunk Control | Change from baseline (Pre-Intervention), after 20 sessions, after 40 sessions, after 60 sessions and after 3 months post 60 sessions(each session is 1.5 hours)
  Participants will be tested in a seated position with arms and back unsupported on a bench with hip and knee both at 90 degrees of flexion and feet supported. Trunk control will be examined with a therapist progressively changing the level of support, starting at the shoulder girdle and axilla to assess cervical (head) control. They will then progress to the inferior-scapula (mid-thoracic), lower-ribs (lower thoracic), below-ribs (upper lumbar), pelvis (lower lumbar) and no support, to measure full trunk control. Pelvis will be placed in a neutral position via manual support for all testing, except for the no support level.
Modified Function Reach (MFR) | Change from baseline (Pre-Intervention), after 20 sessions, after 40 sessions, after 60 sessions and after 3 months post 60 sessions(each session is 1.5 hours)
  Participants will be in a sitting position with hip, knees, and ankles in 90 degrees flexion, with feet flat on the floor. The initial reach will be measured using a yard stick with participant reaching (leaning) as far as possible (front, right, and left). Distance covered, in centimeters from initial position to furthest reaching at the level of the 3rd metacarpal, will be recorded in all 3 directions.

SECONDARY OUTCOMES:
Center of Pressure (CoP) displacement | baseline (Pre-Intervention), After 60 intervention Sessions (each session is 1.5 hours) and 3 months after 60 sessions end
  Center of pressure is the location on the supporting surface where the resultant vertical force vector would act if it could be considered to have a single point of application. A shift of CoP is an indirect measure of postural sway and thus a measure of a person's ability to maintain balance.
Angular Excursions of the Trunk | baseline (Pre-Intervention), After 60 Intervention sessions (each session is 1.5 hours) and 3 months after 60 sessions end
  Degrees of flexion/extension, adduction/abduction and rotation, using wireless motion sensors.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea L Behrman, PT, PhD, Principal Investigator — University of Louisville
Locations (1):
- Kentucky Spinal Cord Injury Res Center, University of Louisville, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No